CLINICAL TRIAL: NCT03472807
Title: An Investigation of Susceptibility Genes for Rare Cancers in Children by Exome Sequencing
Brief Title: EXOme Rare Cancers in Children (EXOCARE)
Acronym: EXOCARE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusions stopped due to lack of inclusions
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-A01833-50
Record Dates: First submitted 2018-01-29; First posted 2018-03-21 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Predisposition, Genetic; Cancer Childhood; Development Delay
MeSH Terms: conditions — Genetic Predisposition to Disease; Neoplasms; Learning Disabilities

STUDY DESIGN:
Intervention Model Description: prospective multicenter study, not therapeutic,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cancer patient (Other): * Collection of blood sample or saliva
  * Collection of a tumor sample taken before the participation of the patient in study
  * Collection of blood sample if tumor sample is not available
  Interventions: Other: Collection of blood sample or saliva; Other: Collection of a tumor sample taken before the participation of the patient in study; Other: Collection of blood sample if tumor sample is not available
- Parent of cancer patient (Other): -Collection of blood sample or saliva
  Interventions: Other: Collection of blood sample or saliva

INTERVENTIONS:
Other: Collection of blood sample or saliva — at Inclusion
Other: Collection of a tumor sample taken before the participation of the patient in study — at Inclusion
  Arms: Cancer patient
Other: Collection of blood sample if tumor sample is not available — at Inclusion
  Arms: Cancer patient

SUMMARY:
Other than high-dose radiation and previous chemotherapy, few strong risk factors have been identified as causes of childhood cancer. Geneticists estimate that 5 to 10% of all cancers diagnosed during the paediatric period occur in children born with a genetic mutation, increasing their lifetime risk of neoplasia. Such genetic risk is higher in children with congenital anomalies and specific genetic syndromes. Some germline genetic alterations are well known (e.g. P53 protein (P53), Neurofibromatosis type 1(NF1)), however many children with none of these mutations have clinical presentations that strongly suggest the involvement of a genetic predisposition. Comprehensive genetic testing for all such patients is an important factor for improving disease surveillance. Such opportunities are now available thanks to whole exome sequencing (WES). In oncology, an important clinical application of WES will be to routinely identify mutations associated with inherited cancer predispositions and to guide cancer risk-management decisions.

Our project is a national translational multicenter genetics study aimed at identifying genes involved in paediatric cancer predisposition by WES in a very select population of children with both developmental delay and cancer. Our project relies on the TED register (Tumeur Et Développement), an initiative by the French organisation SFCE (Société Française de lutte contre les Cancers et les leucémies de l'Enfant et de l'Adolescent) involving 30 child cancer units in France. This database includes the information of more than 500 paediatric cancer patients with congenital abnormalities. The investigators plan to sequence the germline and tumour exome of 100 patients with developmental delay in a trio-design consisting of 300 people and 100 tumours.

The investigators believe that the ExoCaRe project will provide answers to the genetic origins of certain particular childhood cancers. The ExoCaRe project relies on a genetic study to identify genetic risk factors for rare forms of childhood cancer and aims to establish more personalised treatment. It is aimed at improving genetic counselling for families and will be fully integrated in the genetic counselling process. The information provided by our study will be used to improve the management approach to an initial cancer by clarifying the risks of other cancers in related families. The investigators hope to identify new germline genes predisposing to cancer that will be of interest in understanding tumour biology.

DETAILED DESCRIPTION:
-Primary objective : Our aim is to identify new mutations and genes involved in paediatric cancer predisposition associating developmental delay by WES of a sub-cohort of patients included in the TED database.

-Secondary objectives :

1. Describe inherited predisposition to cancer.
2. Improve genetic counselling processes.
3. Initiate clinical exome sequencing in childhood cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* For "Patient cancer" :

  * Child having developed a cancer combined with a delay of development and\or an intellectual deficiency before the age of 18 years and followed for a cancer of the child in one of hospital center of the Société Française de lutte contre les Cancers et les leucémies de l'Enfant et de l'adolescent (SFCE)
  * At least a parent still alive and available to make genetic analyses
* For "Parent of cancer patient" :

  * Parent whose child meets the criteria of inclusion of "Cancer patient"

Exclusion Criteria:

* For "Cancer patient" :

  * Genetic predisposition already identified at the child
  * Absence of histological confirmation
  * Child died without DNA of the available germinal lineage
* For "Parent of cancer patient" :

  * Parent whose child doesn't meets the criteria of inclusion of "Cancer patient"

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Number and type of germline and somatic genetic variants of pathological significance and associated with the disease. | At inclusion
  WES and RNA sequence data will be used to identify and characterise germline and somatic genetic variants of pathological significance and associated with the disease.
  Descriptive statistics, such as counts and proportions of variants of pathological significance risk will be computed within each patient and family.

SECONDARY OUTCOMES:
Related to secondary objectives (1) : Identification of biological pathways involved in childhood cancer predisposition. | At inclusion
  The deleterious mutations that the investigators will identify in genes related to childhood cancer predisposition will help to have a comprehensive framework of biological pathways involved in childhood cancer predisposition.
Related to secondary objectives (2) : Overall success rate. | At inclusion
  Success is defined by the combined successes of quality interpretable genomic data are generated from sequencing tumor and germline tissues, and communicating genomic test results to the primary oncologist and the patient and his/her parents.
Related to secondary objectives (3) : Number of clinical criteria justifying a WES. | At inclusion
  Descriptive statistics, such as counts and proportions of success by clinical presentation of the disease, by cancer types, by features of developmental delay, and, by class of age.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle PELLIER, Pr, Principal Investigator — UH Angers
Locations (27):
- France (26):
  - University Hospital of Amiens, Amiens
  - University Hospital of Angers, Angers
  - Cancer Center Bergonie Institut, Bordeaux
  - University Hospital of Bordeaux, Bordeaux
  - University Hospital of Brest, Brest
  - University Hospital of Clermont Ferrand, Clermont-Ferrand
  - University Hospital of Dijon, Dijon
  - University Hospital of Grenoble, Grenoble
  - University Hospital of Lille, Lille
  - University Hospital of Limoges, Limoges
  - Institut of Haematology and Paediatric Oncology of Lyon, Lyon
  - University Hospital of Marseille, Marseille
  - University Hospital of Montpellier, Montpellier
  - University Hospital of Nancy, Nancy
  - University Hospital of Nantes, Nantes
  - University Hospital of Nice, Nice
  - Institut Curie, Paris
  - University Hospital of Kremlin Bicetre, Paris
  - University Hospital of Necker, Paris
  - University Hospital of Trousseau, Paris
  - University Hospital of Rennes, Rennes
  - University Hospital of Rouen, Rouen
  - University Hospital of Saint Etienne, Saint-Etienne
  - University Hospital of Strasbourg, Strasbourg
  - University Hospital of Tours, Tours
  - Institut Gustave Roussy, Villejuif
- University Hospital of Saint Denis de La Reunion, Saint-Denis, Reunion